CLINICAL TRIAL: NCT07213492
Title: A Bridge to Better Days: A Pilot Study of a Multimodal Intervention to Support the Successful Transition From Hospital to Community Care for People Living With Bipolar Disorder
Brief Title: Multimodal Intervention to Support Hospital-to-Community Transition in Bipolar Disorder
Acronym: BTBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18669
Record Dates: First submitted 2025-09-16; First posted 2025-10-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Bipolar Disorder (BD); Psychosis
Keywords: Bipolar Disorder; Psychoeducation; Insight; Psychosis; Multimodal Intervention; Early-Stage Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-Modal Transitional Care Intervention (Experimental): Participants receive a 6-month structured intervention including: (1) 6 sessions of group-based psychoeducation, (2) biweekly peer support for individuals and families, and (3) two sessions of personalized clinical guidance for community healthcare providers.
  Interventions: Behavioral: Group-Based Psychoeducation; Behavioral: Peer Support; Behavioral: Personalized Support for Community Healthcare Provider

INTERVENTIONS:
Behavioral: Group-Based Psychoeducation — Participants attend a six-session, group-based psychoeducation program delivered over 8 weeks. Sessions focus on improving insight into bipolar disorder, relapse prevention, lifestyle strategies (e.g., sleep, nutrition, substance use), and digital literacy. The aim is to enhance understanding of illness and support long-term functioning.
Behavioral: Peer Support — Trained peer support workers provide biweekly sessions over 6 months to participants. The sessions are based on the CANMAT/ISBD Patient and Family Guide and include emotional support, psychoeducation, and shared experience. Each participant receives up to 12 sessions aimed at improving engagement and understanding of illness.
Behavioral: Personalized Support for Community Healthcare Provider — The research team provides two personalized support sessions over 6 months to each participant's healthcare provider (e.g., family doctor or psychiatrist). Support includes treatment recommendations based on the CANMAT/ISBD 2018 Guidelines and training on the C-IMPACT BD web-based clinical decision support tool.

SUMMARY:
People with bipolar disorder (BD) are at high risk of relapse following hospital discharge, partly due to a lack of BD-specific expertise and resources within community services required for comprehensive treatment. Although clinical guidelines recommend combining medication and psychosocial support, and research shows that early intervention is associated with improved outcomes, no structured care programs currently exist for individuals in the early stages of BD, contributing to chronic illness progression and preventable hospitalizations. This open-label pilot trial will assess the feasibility, acceptability, and preliminary effectiveness of a structured care pathway to support the transition from hospital to community care. The intervention includes group-based psychoeducation, individual peer support, and personalized support for community healthcare providers to improve illness insight, treatment adherence, and symptom management.

DETAILED DESCRIPTION:
This is a 6-month, open-label pilot study of the feasibility, acceptability, and preliminary effectiveness of a multimodal transitional-care intervention for individuals with BD who have recently been discharged from the hospital. The intervention comprises a brief group psychoeducation program (6 clinician-facilitated sessions delivered over up to 8 weeks), individualized peer support (biweekly one-on-one sessions for ~12 total across 6 months), and optional personalized support for participants' primary healthcare providers (two collaborative sessions over 6 months offering guideline-based recommendations and access/training to a clinical decision-support app). Ten patient-participants who meet the inclusion criteria will be enrolled over 6 months; this sample will be used to estimate recruitment, retention, adherence, satisfaction, and safety parameters, and to inform power and procedures for a subsequent randomized controlled trial. Participants will be recruited from St. Joseph's Healthcare Hamilton (SJHH) outpatient clinics, the community and the ENABLE research registry at SJHH (Hamilton, ON, Canada). Eligible adults are 18-35 years old with a BD diagnosis within the past 24 months and a history of psychosis and/or limited illness insight; all must meet inclusion/exclusion criteria and provide written informed consent. After obtaining consent, eligibility will be confirmed with the Mini-International Neuropsychiatric Interview (MINI) and the Mood Disorders Insight Scale (MDIS). Study visits occur at three timepoints: baseline, post-psychoeducation, and post-multimodal intervention (6 months). At each assessment time point, clinicians and/or patient-participants will complete validated measures; socio-demographic and clinical history will be collected at baseline. Feasibility will be assessed through recruitment, enrollment, adherence (session attendance/completion), and retention metrics; acceptability through patient-participant and healthcare-provider satisfaction questionnaires; and safety through prospective monitoring of emergent symptoms, acute relapse, emergency visits, hospitalizations, and suicide-related events. Data will be summarized primarily with descriptive statistics (means, standard deviations, frequencies); exploratory pre-post comparisons (e.g., t-tests or chi-square) will evaluate the signal of change in symptoms, insight, functioning, lifestyle, and quality of life. The results of this study will determine whether delivering a structured psychoeducation + peer-support + provider-support care pathway during the transition from hospital to community is feasible and acceptable for early-stage BD, and will guide sample-size calculations, procedures, and implementation strategies for a subsequent randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patient-participants must be between 18 and 35 years old.
* Diagnosis: Must have been diagnosed with bipolar disorder within the past 24 months.
* Clinical Features: Must have experienced psychosis and/or a lack of insight into their illness at the time of enrollment.
* Language Proficiency: Must be able to understand and speak English.

Exclusion Criteria:

* Severe Psychiatric Conditions: Individuals with a severe psychiatric condition that would prevent them from safely engaging in the intervention.
* Cognitive or Medical Impairment: Those with significant cognitive impairment or a medical condition that interferes with their ability to participate in psychoeducation or peer-support sessions.
* Substance Use Disorder: Individuals with an active substance use disorder that may impact adherence to the intervention.
* Language Barriers: Participants who do not speak English and are unable to engage in study sessions without language support.
* Concurrent Participation in Similar Programs: Individuals who are already enrolled in another structured psychoeducational or peer-support program that could interfere with study outcomes.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Multi-Modal Transitional Care Intervention | From enrollment to the end of intervention at 6 months.
  Feasibility will be assessed using three descriptive indicators: 1) Recruitment rate: the proportion of eligible patient-participants and community healthcare providers who consent to participate. 2) Retention rate: the proportion of enrolled participants who remain in the study until the final follow-up. 3) Intervention adherence: participant adherence to each intervention component, including the number of sessions attended and number of dropouts.
  Each indicator will be analyzed separately to determine the feasibility of implementing the multi-modal transitional care intervention.
Acceptability of the Multi-Modal Transitional Care Intervention | Administered at the end of the intervention (Month 6).
  Acceptability will be measured using post-intervention surveys completed by patient-participants and community healthcare providers. Surveys will assess satisfaction and perceived usefulness of the intervention using Likert-scale items, with the option to provide additional information via open-ended questions.

SECONDARY OUTCOMES:
Change in Depression Symptoms (MADRS) | Baseline and Month 6 (end of intervention).
  Clinician-rated 10-item scale assessing depressive symptoms over the past 7 days. Items are rated on a 7-point Likert scale, with higher scores indicating more severe symptoms.
Change in Mania Symptoms (YMRS) | Baseline and Month 6 (end of intervention).
  Clinician-rated 11-item scale assessing manic symptoms using clinical interview and observation. Items scored 0-4 or 0-8, with higher scores indicating more severe mania.
Change in Anxiety Symptoms (GAD-7) | Baseline, Mid-intervention (Month 3), and Month 6 (end of intervention).
  7-item self-report scale assessing anxiety over the past 2 weeks. Items scored 0-3; higher scores reflect greater anxiety.
Change in Depression Severity (Patient Health Questionnaire) (PHQ-9) | Baseline, Mid-intervention (Month 3), and Month 6 (end of intervention).
  9-item self-report scale evaluating the presence and severity of depression symptoms over the past 2 weeks. Each item scored 0-3; higher scores indicate greater severity.
Change in Insight (MDIS) | Baseline and Month 6 (end of intervention).
  Self-report scale assessing insight in mood disorders. Participants respond "Agree," "Disagree," or "Unsure." Higher scores indicate better insight.
Change in Psychosocial Functioning (FAST) | Baseline and Month 6 (end of intervention).
  Clinician-administered scale assessing functioning across six domains (autonomy, work, cognition, finances, relationships, leisure). Each item rated 0-3.
Change in Cognitive Complaints (COBRA) | Baseline and Month 6 (end of intervention).
  16-item self-report questionnaire measuring cognitive dysfunction in bipolar disorder. Each item scored 0-3; higher scores indicate more impairment.
Change in Quality of Life (Q-LES-Q-SF) | Baseline, Mid-intervention (Month 3), and Month 6 (end of intervention).
  16-item self-report scale assessing satisfaction and enjoyment in multiple life areas over the past week. Items rated on a 5-point scale.
Change in Lifestyle Behaviours (SMILE) | Baseline and Month 6 (end of intervention).
  Self-report scale measuring behaviours across seven lifestyle domains (diet and nutrition, substance use, physical activity, stress management, restorative sleep, social support, and environmental exposures). Items scored on a 4-point scale; higher scores reflect healthier lifestyle.

OTHER OUTCOMES:
Safety Monitoring: Relapse, Hospitalization, and Risk | Throughout the 6-month intervention period.
  Monitoring and documentation of adverse events including psychiatric relapse, hospitalizations, and suicide attempts throughout the intervention period.
Sociodemographic Factors | Baseline and Month 6 (end of intervention).
  Demographic and clinical background data will be collected, including gender, age, ethnicity, marital status, education level, income, medical and psychiatric history, family history of psychiatric disorders, medication usage, and treatment history.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Currently, we do not have the plan of individual participant data (IPD) sharing.

REFERENCES:
- [Background] Yatham LN, Kennedy SH, Parikh SV, Schaffer A, Bond DJ, Frey BN, Sharma V, Goldstein BI, Rej S, Beaulieu S, Alda M, MacQueen G, Milev RV, Ravindran A, O'Donovan C, McIntosh D, Lam RW, Vazquez G, Kapczinski F, McIntyre RS, Kozicky J, Kanba S, Lafer B, Suppes T, Calabrese JR, Vieta E, Malhi G, Post RM, Berk M. Canadian Network for Mood and Anxiety Treatments (CANMAT) and International Society for Bipolar Disorders (ISBD) 2018 guidelines for the management of patients with bipolar disorder. Bipolar Disord. 2018 Mar;20(2):97-170. doi: 10.1111/bdi.12609. Epub 2018 Mar 14. PMID 29536616
- [Background] Gomes FA, Dumay H, Fagen J, Palma N, Milev R, Brietzke E. Does the Ranking Matter? A Retrospective Cohort Study Investigating the Impact of the 2018 CANMAT and ISBD Guidelines for the Management of Patients with Bipolar Disorder Treatment Recommendations for Acute Mania on Rehospitalization Rates. Can J Psychiatry. 2023 Aug;68(8):605-612. doi: 10.1177/07067437231156235. Epub 2023 Feb 21. PMID 37551100
- [Background] Correll CU, Galling B, Pawar A, Krivko A, Bonetto C, Ruggeri M, Craig TJ, Nordentoft M, Srihari VH, Guloksuz S, Hui CLM, Chen EYH, Valencia M, Juarez F, Robinson DG, Schooler NR, Brunette MF, Mueser KT, Rosenheck RA, Marcy P, Addington J, Estroff SE, Robinson J, Penn D, Severe JB, Kane JM. Comparison of Early Intervention Services vs Treatment as Usual for Early-Phase Psychosis: A Systematic Review, Meta-analysis, and Meta-regression. JAMA Psychiatry. 2018 Jun 1;75(6):555-565. doi: 10.1001/jamapsychiatry.2018.0623. PMID 29800949
- [Background] Simjanoski M, de Azevedo Cardoso T, Frey BN, Minuzzi L, De Boni RB, Balanza-Martinez V, Kapczinski F. Lifestyle in bipolar disorder: A cross-sectional study. Span J Psychiatry Ment Health. 2023 Oct-Dec;16(4):244-250. doi: 10.1016/j.rpsm.2023.04.001. Epub 2023 May 26. PMID 37839960
- [Background] Ratheesh A, Hett D, Ramain J, Wong E, Berk L, Conus P, Fristad MA, Goldstein T, Hillegers M, Jauhar S, Kessing LV, Miklowitz DJ, Murray G, Scott J, Tohen M, Yatham LN, Young AH, Berk M, Marwaha S. A systematic review of interventions in the early course of bipolar disorder I or II: a report of the International Society for Bipolar Disorders Taskforce on early intervention. Int J Bipolar Disord. 2023 Jan 3;11(1):1. doi: 10.1186/s40345-022-00275-3. PMID 36595095